CLINICAL TRIAL: NCT04432805
Title: Descriptive and Evaluation Study of the Use of Pulmonary Ultrasound in the Initial Management of Pregnant Women in the Context of COVID-19
Acronym: LUSCOVIDPREG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-30; 2020-A01303-36 (Other: ID RCB)
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Pregnant Women Suspected of COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Experimental): Pregnant women suspected of COVID-19
  Interventions: Device: Performing of lung ultrasound

INTERVENTIONS:
Device: Performing of lung ultrasound — Performing of lung ultrasound at bedside in labor ward or in COVID unit

SUMMARY:
Cohort prospective study.

Objectives :

Primary objective:

To describe the lung ultrasound lesions in pregnant women in case of suspected or confirmed COVID-19

Secondary objectives:

* To compare the lung ultrasound lesions with chest Computed Tomography -scanner (CT-Scan) lesions
* To evaluate the performances of the lung ultrasound to diagnose COVID-19 in pregnant women
* To evaluate predictive value of different lung ultrasound lesions for intensive care unit admission of pregnant women with suspected or confirmed COVID-19
* To describe the pregnancy issues of the study population

Course of the study:

* Inclusion of pregnant suspected of having COVID-19 and cared following the service protocol
* Performing of lung ultrasound at bedside in labor ward or in COVID unit

Primary outcome:

Lung ultrasound lesions (and corresponding score) at the moment of the initial management of pregnant women suspected or confirmed with COVID-19 (having a nasopharyngeal Reverse Transcription Polymerase Chain Reaction (RT-PCR) SARS-CoV-2 and a chest CT-scan)

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Gestational age greater than or equal to 22 weeks of gestation
* Pregnant women suspected of COVID-19 :
* already having a nasopharyngeal RT-PCR for the SARS-CoV-2
* AND having a chest CT-scan or waiting for this exam
* Women giving a writing consent to participate

Exclusion Criteria:

* Women giving an opposition to participate
* Women not enough fluent in French to benefit from clear and intelligible information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Description of the lesions | 4 months
  Description of the lesions in each of the 6 pulmonary quadrants on the right and left. Establishment of the ultrasound score corresponding to the sum of the scores attributed to each type of lesion in each quadrant (0: normal, 1: spaced comet tails, 2: curtain comet tails, 3: consolidation).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No